CLINICAL TRIAL: NCT02078583
Title: The Effect of Analgesia Based Sedation Protocol on Brain Function of Critical Care Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEKING SEDATION
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Fentanyl; Remifentanil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Remifentanil，midazolam (Experimental): Remifentanil 1µg/kg/hr intravenous pump and Midazolam loading dose 0.05mg/kg followed by 0.02~0.1mg/kg/h continuous intravenous pump for 7days or extubation
  Interventions: Drug: Remifentanil
- Fentanyl，midazolam (Experimental): Fentanyl 1µg/kg/hr intravenous pump and Midazolam loading dose 0.05mg/kg followed by 0.02~0.1mg/kg/h continuous intravenous pump for 7days or extubation
  Interventions: Drug: Fentanyl
- Normal saline (Placebo Comparator): Normal saline1µg/kg/hr intravenous pump and Midazolam loading dose 0.05mg/kg followed by 0.02~0.1mg/kg/h continuous intravenous pump for 7days or extubation
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Fentanyl
  Arms: Fentanyl，midazolam
Drug: Remifentanil
  Arms: Remifentanil，midazolam
Drug: Normal saline
  Arms: Normal saline

SUMMARY:
Benzodiazepines is a commonly uesd sedative medication,there are many reports that Benzodiazepines is associated with delirium ,but using of analgesia reduces benzodiazepines requirements .The purpose of this study is to determine whether analgesia based sedation protocol reduces the incident of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Signing a consent form
* postoperative patient
* Requirement for mechanical ventilation and anticipate time of mechanical ventilation more than 24 hours
* Requirement for sedation
* Age more than 18 and less than 85 years old

Exclusion Criteria:

* Unstable blood circulation
* Heart rate less than 50 beats per minute
* II ° ～ III ° atrioventricular conduct block
* Intracranial lesions 、neurosurgical intervention and mental disability inability to cooperate;
* Receipt of antipsychotics 、hypnotic drugs before surgery ;
* Alcohol abuse;
* Liver failure class Child-Pugh C;
* Acute Respiratory Distress Syndrome;
* Acute or chronic renal failure;
* Other severe diseases ,septic shock;
* Receipt of neuromuscular blocking drug;
* Pregnancy and nursing woman;
* Allergy to investigational drug or other contraindication.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The incidence and duration of delirium in patients with different regimens | 1 day

SECONDARY OUTCOMES:
Mortality | 28 days
Ventilator-free days | an expected average of 7 days
Mean days of mechanical ventilation | an expected average of 7 days
Length of ICU stay | an expected average of 7 days
Index of anesthesia depth monitoring | From admission to ICU to weaning,about 7 days
  Analgesic level、sedation level、brain function、 blood perfusion for peripheral and brain circulation、sleep stages and variation of blood volume
Infusion velocity and total dose of sedative drugs in different groups | From admission to ICU to extubation or drug withdrawal,about 7 days
Plasma melatonin level | Every 6 hours during the next ICU day
Total rescue dose of midazolam | Seven days after giving midazolam to patient
Variations of HR、RR、BP、SpO2 | an expected average of 7 days